CLINICAL TRIAL: NCT05739006
Title: A Multicenter, Double-Blind, Randomized Clinical Study to Evaluate the Pharmacokinetics and Safety of BCD-201 (JSC BIOCAD, Russia) and Keytruda® in Patients With Different Advanced Malignancies
Brief Title: Clinical Trial to Evaluate the PK and Safety of BCD-201 and Keytruda® in Patients With Advanced Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-201-1
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Melanoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): BCD-201 200 mg by intravenous infusions once every 3 weeks
  Interventions: Drug: BCD-201
- Group 2 (Active Comparator): Keytruda 200 mg by intravenous infusions once every 3 weeks
  Interventions: Drug: Keytruda

INTERVENTIONS:
Drug: BCD-201 — up to 8 treatment cycles
  Other Names: pembrolizumab
  Arms: Group 1
Drug: Keytruda — up to 8 treatment cycles
  Other Names: pembrolizumab
  Arms: Group 2

SUMMARY:
Clinical study BCD-201-1 is a double-blind randomized study of the pharmacokinetics (PK), pharmacodynamics (PD), safety, and immunogenicity of BCD-201 versus Keytruda following intravenous administration to subjects with advanced unresectable, metastatic, or recurrent melanoma and NSCLC.

The study aimed to establish the equivalence of PK and similarity of the safety, immunogenicity, and PD profiles of BCD-201 and Keytruda.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Body weight 60 to 90 kg;
* Histologically confirmed melanoma or NSCLC (patients with NSCLC are eligible to participate if high tumor PD-L1 expression [≥50%] is confirmed by local or central laboratory results);
* ECOG score 0-1;
* Laboratory test results consistent with adequate functioning of systems and organs;
* Willingness of males and females of childbearing potential to use highly effective contraceptive methods from the signing of the informed consent form, throughout the study and within 6 months after the administration of the last product dose

Exclusion Criteria:

* Indications for radical therapy (surgery, radiation therapy);
* Previous systemic anti-tumor therapy for advanced unresectable, recurrent or metastatic melanoma or NSCLC (history of neoadjuvant or adjuvant therapy is acceptable provided that the treatment was completed at least 6 weeks prior to randomization);
* Active metastases in the central nervous system and/or carcinomatous meningitis;
* Patients with severe concomitant disorders, life-threatening acute complications of the primary disease (including massive pleural, pericardial, or peritoneal effusions requiring intervention, pulmonary lymphangitis, bleeding or organ perforation) at the time of signing the informed consent and during the screening period;
* For patients with NSCLC: presence of activating EGFR mutations/ALK translocations;
* Concomitant diseases and/or conditions that significantly increase the risk of AEs during the study;
* Active, known or suspected autoimmune disorders (subjects with type 1 diabetes mellitus or hypothyroidism requiring only hormone-replacement therapy and those with skin disorders [vitiligo, alopecia, or psoriasis] not requiring systemic therapy are eligible to participate);
* The need for therapy with glucocorticoids or any other drugs with immunosuppressive effects within 14 days prior to randomization;
* History of (non-infectious) pneumonitis requiring glucocorticoid therapy or pneumonitis at the time of screening;
* Hypersensitivity or allergy to any of the pembrolizumab product components;
* Pregnancy or breastfeeding, as well as intention to become pregnant or father a child during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
AUC(0-504) of pembrolizumab | pre-dose to week 25, 77 timepoints
  area under the drug concentration-time curve in the time interval from 0 to 504 hours

SECONDARY OUTCOMES:
AUC(0-∞) of pembrolizumab | pre-dose to week 25, 77 timepoints
  Area under the drug concentration-time curve in the time interval from 0 to ∞
Cmax | pre-dose to week 25, 77 timepoints
  maximum concentration of pembrolizumab
Tmax | pre-dose to week 25, 77 timepoints
  time to maximum concentration of pembrolizumab
T½ | pre-dose to week 25, 77 timepoints
  Half-life period
Vd | pre-dose to week 25, 77 timepoints
  Steady-state volume of distribution of the drug substance
Cmin | pre-dose to week 25, 77 timepoints
  minimum concentration of pembrolizumab
kel | pre-dose to week 25, 77 timepoints
  Elimination rate constant
Cl | pre-dose to week 25, 77 timepoints
  Total clearance
Safety assessment | Day 1 to Day 169
  proportion of patients with any adverse events (AEs); • proportion of patients with severe AEs; proportion of patients who discontinued study therapy due to AEs; • proportion of patients with immune-mediated AEs
Immunogenicity assessment | pre-dose to week 25, 5 timepoints
  the frequency of binding and neutralizing anti-pembrolizumab antibody production
To compare the results of pilot assessment of BCD-201 and Keytruda efficacy | Day 1 to week 25
  overall response rate (ORR)

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - "Russian Cancer Research Center named after N.N. Blokhin "of the Ministry of Health of the Russian Federation, Moscow
  - Budgetary healthcare institution of the Omsk region "Clinical oncological dispensary", Omsk
  - State Budgetary Healthcare Institution "Saint Petersburg Clinical Research and Practice Center for Specialized Medical Care (Oncology)", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No